CLINICAL TRIAL: NCT04520282
Title: Haemostatic Variables in Snakebite: a Regional Prospective Cohort to Identify the Role of Global Coagulation Assays and Serial Laboratory Testing in the Management of Snakebite Coagulopathy
Brief Title: Hemostatic Variables In Snakebite Study
Acronym: HISS
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Siju V Abraham, MD, Associate Professor, Jubilee Mission Medical College and Research Institute
Other Study IDs: 01/20/IEC/JMMC&RI; U1111-1252-7998 (Other: World Health Organisation)
Record Dates: First submitted 2020-05-31; First posted 2020-08-20 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Snake Bites; Coagulopathy, Consumption
Keywords: global coagulation assay; hemostatic variables; coagulopathy; VICC; DIC; Venom induced consumptive coagulopathy; Disseminated intravascular coagulation; ROTEM; CWA; clot waveform analysis; 20'WBCT; Clotting time; thromboelastometry; viscoelastometry; blood cell indices; snakebite; hematotoxic
MeSH Terms: conditions — Snake Bites; Disseminated Intravascular Coagulation; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background

Novelty The global assays of coagulation, namely the viscoelastometric tests and clot waveform has never been studied in detail before in snakebite victims.

The pathophysiology of VICC including specific factor deficiencies and serial trend in blood cell indices amongst various hematotoxic snakebite in the region is not known.

No Indian study to date has systematically examined the changes in early laboratory tests results in envenomed and non envenomed snakebite victims.

DETAILED DESCRIPTION:
The problem:

Snakebite is a neglected disease of the poor in India. Nearly 50,000 individuals die of snake bite every year in the country, making it the region with most number of snakebite related deaths in the world.

Snakebite though is one of the leading cause of mortality and morbidity globally, it is in fact a "local" problem which warrants a regionalized approach. The venom characteristics of snakes and their response to treatment vary across geographical regions, even within the same species.

Therefore the venom sourcing for antivenom production, to clinical characterization of snakebites needs to be regionalized.

Clinical profiling of snakebite has been done in many observational studies across the region but a comprehensive prospective regional profiling of laboratory parameters including the global assays have not been done to date.

The health care in India is mostly out of one's own pocket, and the victims are of the lower socio economic strata the health care costs are seldom affordable. Research in the field is also sparse due to lack of funding for the same. The investigators through this research aim to study the clinical and laboratory profile of snakebite victims presenting to a tertiary care snakebite treatment centre in central Kerala and the role of global coagulation assays in the management of the same.

Once answered, the research question, would provide a better understanding of the hematotoxic snakebite in the region.

It could aid in better patient care strategies, including possible determination of a better test for coagulopathy, judicious antivenom and blood product usage.

Its relevance in local, national and international context:.

Snakebite being region specific warrants a region specific approach to the problem. Venomous species like Humpnosed pit viper (Hypnale hypnale) envenomation which is the second most common snakebite (first being Daboia russelli ) in the region is a serious problem that needs better understanding.

This would be a model which can be replicated in selected tertiary care snakebite centers across the country. Answering these research questions across the country would lead to better understanding of coagulopathy in snakebite, its response to antivenom and blood products in India.

It may also lead to quantifying the need for region specific antivenom in the country.

No Indian study has systematically examined the changes in early laboratory tests results in envenomed and non envenomed snakebite victims to date.

With the exception of a few case reports there has been no studies that has looked at the performance of global coagulation assays in the country.

The country that becomes the largest contributor of global burden of snake bite in terms of mortality is India.

This model if applicable in India, should be replicable elsewhere too. Ten years back, the investigators would not have been able to envision this study, since the understanding of the process of snake bite related coagulopathy was limited, and it was national projects like the Australian snake bite project implemented elsewhere that form the basis for the current understanding of the problem of snakebite.

In the international context many other low and middle income countries that are burdened by snake bites would benefit from any result in terms of a better bedside coagulation test (like CWA or MLW) or a cheaper blood indices (DNI) to prognosticate snake envenomation.

The understanding of coagulopathy in snakebite is now changing. Conventionally, although this coagulopathy is likened to disseminated intravascular coagulation (DIC), in the recent years, it has been described as venom-induced consumptive coagulopathy (VICC).

VICC defers from DIC in its rapidity of both onset and resolution. It used to be compared to Disseminated Intravascular Coagulation, but now the understanding of the same is changing and more recently the term VICC- Venom induced consumptive coagulopathy has been introduced. The snake venom in India are known to contain Factor V activators (D russelli), Factor X activators (D russelli), prothrombin activators (PTA) (Echis sp.), thrombin like enzymes (TLE) and fibrinogenases (Trimeresurus sp,. Hypnale hypnale). The above mentioned findings are mostly from studies in Srilanka, with assays done in samples frozen and sent to Australia, by the same team of investigators.

There are not many properly conducted study from any region of India that helps understand the pathophysiology better.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with history suggestive of snakebite presenting within 6 hours of snakebite AND
2. All providing a written informed consent and/or assent

Exclusion Criteria:

1. All patients of stings or bites other than snakes
2. All patients who received antivenom or blood products at another institute
3. All patients with known hematological malignancies, coagulation disorders, chronic liver or renal failure.
4. All patients known to be on warfarin, heparin or any newer oral or injectable anticoagulants
5. All withdrawing a consent later on, or withdrawing assent later on-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with history suggestive of snakebite presenting within 6 hours of snakebite and providing a written informed consent and/or assent would be included in the study
  Definitions:
  'Snakebite' OR 'History suggestive of snakebite' would be defined as, patients or their bystander claiming in sound mind not and not under the influence of any inebriants, to have witnessed being bitten by a snake, OR, patient with clinical features of snakebite as suspected by the clinician on floor
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
To study the serial change in CT of snakebite victims | up to 30 days
  Change from baseline (sample taken at admission) for clotting time would be recorded in minutes and seconds assessed at 1 hour (post admission), 1 hour 30 mins (post admission), 3 hours (post admission), 6 hours (post bite), 6 hours post antivenom, 6 hours after blood products or 12 hours after antivenom and at discharge or at 30 days (whichever is earlier)
To study the serial change in fibrinogen levels of snakebite victims | up to 30 days
  The change in fibrinogen levels from baseline (sample taken at admission, 0 hour), 6 hour post bite, 6 hours post antivenom,12 hours post antivenom, 6 hours after blood products and at discharge or at 30 days (whichever occurs earlier), measured in weight per volume (milligram per decilitre).
To study the serial change in D dimer levels of snakebite victims | up to 30 days
  The change D dimer from baseline (sample taken at admission, 0 hour), 6 hour post bite, 6 hours post antivenom,12 hours post antivenom, 6 hours after blood products and at discharge or at 30 days (whichever occurs earlier) measured in weight per volume ( micrograms per decilitre respectively).

SECONDARY OUTCOMES:
Diagnostic accuracy of Clotting Time in detecting coagulopathy | 48 hours
  Sensitivity and specificity of Clotting Time (minutes) done using Modified Lee and White method (MLW) in detecting coagulopathy compared to conventional coagulation test (PT, aPTT)
Diagnostic accuracy of 20'WBCT, MLW, Delayed reading of 20'WBCT in detecting coagulopathy | 48 hours
  Sensitivity, specificity of
  1. 20'WBCT (minutes)
  2. Delayed reading of 20'WBCT (30'WBCT) in detecting coagulopathy compared to conventional coagulation test (PT, aPTT)
Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of the bedside coagulation tests. | 48 hours
  Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of bedside coagulation tests (20'WBCT, MLW Clotting time, Delayed reading of 20'WBCT, Activated Clotting Time) (before and after antivenom)
Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation conventional coagulation tests | 48 hours
  Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of conventional coagulation tests PT/INR and aPTT (before and after antivenom)
To study the serial change in PT and aPTT-clot waveform of snakebite victims | up to 7 days
  The change of PT and aPTT-clot waveform from baseline (sample taken at admission; 0 Hours) would be recorded in milli absorption (mabs) per second, 6 hours (post bite), 6 hours post antivenom, 12 hours post antivenom ,6 hours after blood products and at discharge or 7 days whichever is earlier
To describe the clinical characteristics of snakebite victims measured as per a pre set proforma | up to 30 days
  The clinical characteristics of snakebite victims, including systemic manifestation and local manifestations would be measured as per a pre set proforma

OTHER OUTCOMES:
Time to envenomation in hematotoxic snakebites in the region | 7 days
  time taken from snakebite, to development of signs or symptoms suggestive of envenomation in the first 7 days post bite measured in days, hours and minutes
Time to envenomation in Russells viper snake bite in the region | 48 hours
  time taken from snakebite, to development of signs or symptoms suggestive of envenomation in the event of a Russells viper (Daboia russellii) bite measured in hours and minutes
Time to envenomation in pitviper (crotaline) snake bite in the region | 48 hours
  time taken from snakebite, to development of signs or symptoms suggestive of envenomation in the event of a pit viper bite Crotaline snakes, like humpnosed pitviper, large scaled pitviper, green pit viper and horseshoe pitviper measured in hours and minutes
To study the serial change in ROTEM waveform of snakebite victims | up to 7 days
  The change in ROTEM waveform would be recorded from baseline (sample taken at admission; 0 Hours) in amplitude (mm) per time (minutes), 6 hours, 6 hours post antivenom,12 hours post antivenom, 6 hours after blood products and thereafter every 6th hourly upto seven days.
To study the serial change in PT, aPTT of snakebite victims | up to 30 days
  Change from baseline (sample taken at admission) for prothrombin time, activated partial thromboplastin time would be recorded in minutes and seconds assessed 6 hours (post bite), 6 hours post antivenom, 6 hours after blood products or 12 hours after antivenom and at discharge or at 30 days (whichever is earlier)
To study the serial change in coagulation factor assays of snakebite victims | up to 7 days
  The change of coagulation factor assays from baseline (sample taken at admission; 0 Hours) would be recorded in international units (IU) per volume (millilitre, decilitre) and at 12 hours post antivenom.
Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of coagulation factor assays. | 48 hours
  Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of coagulation factor assays (before and after antivenom)
Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of Clot Waveform analysis (CWA) and Rotational Thromobelastometry | 48 hours
  Change in coagulopathy in snakebite victims, after antivenom administration as measured by normalisation of the waveforms in CWA and ROTEM (before and after antivenom)
To study the serial change in myoglobin levels of snakebite victims | 7 days
  The change serum myoglobin from baseline (sample taken at admission, 0 hour), 6 hour post bite, 6 hours post antivenom,12 hours post antivenom, 6 hours after blood products and at discharge or at 7 days (whichever occurs earlier) measured in weight per volume ( nanogram per millitre respectively).
To study the correlation of admission proteinuria and incidence of renal failure in 30 days | up to 7 days
  To study the correlation of proteinuria measured using urine dipstick, within 6 hours of envenomation with development of acute kidney injury measured as per RIFLE criteria, within 30 days
To describe the peripheral smear changes in hematotoxic snakebite victims | up to 7 days
  To qualitatively describe the peripheral smear from baseline (sample taken at admission, 0 hour), with 6 hour post bite, 6 hours post antivenom,12 hours post antivenom, 6 hours after blood products and at discharge or at 7 days (whichever occurs earlier)

CONTACTS AND LOCATIONS:
Overall Officials: Siju V Abraham, M D, Principal Investigator — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abraham SV, Rafi AM, Krishnan SV, Palatty BU, Innah SJ, Johny J, Varghese S. Utility of Clot Waveform Analysis in Russell's Viper Bite Victims with Hematotoxicity. J Emerg Trauma Shock. 2018 Jul-Sep;11(3):211-216. doi: 10.4103/JETS.JETS_43_17. PMID 30429630